CLINICAL TRIAL: NCT00874471
Title: Uveitis Gene-Expression Profiling
Status: Completed | Type: Observational
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jim Rosenbaum, Professor, Oregon Health and Science University
Other Study IDs: R01EY015858 (NIH)
Record Dates: First submitted 2009-04-01; First posted 2009-04-02 (Estimated); Last update posted 2014-04-09 (Estimated); Status verified 2014-04

CONDITIONS: Uveitis
MeSH Terms: conditions — Uveitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (10):
- sarcoidosis
- ankylosing spondylitis
- Behcet's disease
- toxoplasmosis
- herpetic acute retinal necrosis
- idiopathic uveitis
- ankylosing spondylitis (no uveitis)
- sarcoidosis (no uveitis)
- Behcet's disease (no uveitis)
- normal control

SUMMARY:
Uveitis is a group of troublesome diseases that collectively represent a cause of blindness comparable to diabetes. Most forms of uveitis are either infectious or immune-mediated. The investigators propose to create a data base on peripheral blood gene expression for patients with 3 of the most important diseases associated with uveitis: ankylosing spondylitis, sarcoidosis, and Behcet's disease. The investigators will quantitatively measure the expression of consistent alteration in peripheral blood from patients with more than 40,000 gene sequences using microarray gene chip technology. This approach is known to detect systemic immune-mediated disease. The investigators will use this data base to:

1. Determine if patients with uveitis and ankylosing spondylitis, sarcoidosis, or Behcet's can be distinguished from a normal population or controls with the same systemic disease but no history of uveitis
2. Determine if the profile of gene expression can distinguish infectious or idiopathic forms of uveitis from patients with spondylitis, sarcoidosis, or Behcet's
3. Determine how this gene profile changes over time as episodic disease such as spondylitis or Behcet's activates or remits
4. Correlate the changes in gene expression with the prognosis of the ocular inflammatory process.

The creation of a gene expression data base for patients with uveitis has the potential to clarify the pathogenesis of disease, establish new diagnostic tools, and provide a means for predicting prognosis.

ELIGIBILITY:
Inclusion Criteria:

* The study group will include patients aged 21 years or older attending the Uveitis Clinic at the Casey Eye Institute at OHSU who have uveitis of the following subtypes:

  1. ankylosing spondylitis
  2. sarcoidosis
  3. Behçet's disease
  4. toxoplasmosis
  5. herpetic acute retinal necrosis; AND
  6. idiopathic uveitis
* Another group of patients, also aged 21 years or more, with the following diseases but no uveitis, will be recruited from the Rheumatology Clinic at OHSU as follows:

  1. ankylosing spondylitis
  2. sarcoidosis; AND
  3. Behçet's disease
* The study group will also include 30 normal control volunteers aged 21 years or older.

Exclusion Criteria:

* Special/vulnerable subject populations (e.g., mentally impaired persons and children) will not be enrolled.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals suffering from selected subtypes of uveitis, individuals suffering from selected autoimmune disease and healthy individuals.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Actual)
Dates: Start 2005-06; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Correlation of blood transcriptome with form of uveitis | time of office visit for disease evaluation

CONTACTS AND LOCATIONS:
Overall Officials: James Rosenbaum, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States